CLINICAL TRIAL: NCT02111148
Title: Urea and Creatinine Versus Nitrazine Test in Vaginal Fluid Wash in Diagnosed Pre Labour Rupture of Membranes
Brief Title: Vaginal Fluid Wash in Pre-labour Rupture of Membranes
Acronym: PROM
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Beni-Suef University (Other)
Collaborators: Cairo University (Other)
Responsible Party: Principal Investigator, Nesreen Abdel Fattah Abdullah Shehata, Beni-Suef University, Beni-Suef University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Diagnostic
Other Study IDs: Beni-Suef 2
Record Dates: First submitted 2014-04-02; First posted 2014-04-11 (Estimated); Last update posted 2021-02-16 (Actual); Status verified 2021-02

CONDITIONS: Disorder of Amniotic Cavity and/or Membrane
Keywords: rupture of membranes, nitrazine, urea, creatinine
MeSH Terms: interventions — Urea; Creatinine; nitrazine yellow; Sodium Chloride

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (3):
- urea and creatinine (Active Comparator): urea and creatinine detected in vaginal fluid wash after injecting of 5 ml saline intavaginally
  Interventions: Procedure: Urea and creatinine
- Nitrazine (Active Comparator): Biochemical description of Nitrazine in the vaginal wash
  Interventions: Procedure: Nitrazine
- saline (Active Comparator): 5ml saline will be injected in vagina of each patient in both groups within 24 hours of membrane rupture.
  Interventions: Drug: 5ml saline

INTERVENTIONS:
Procedure: Urea and creatinine — the vagina will be washed with 5ml saline, urea and creatinine will be detected biochemically in the vaginal wash.
  Arms: urea and creatinine
Procedure: Nitrazine — Nitrazine detection in vaginal wash
  Arms: Nitrazine
Drug: 5ml saline — the vagina will be washed with 5ml saline and vaginal wash will be collected.
  Arms: saline

SUMMARY:
The investigators assess in this study the sensitivity of Urea and Creatinine and that of Nitrazine test in vaginal wash after injecting saline in the vagina of patients with pre-labour rupture of membranes

DETAILED DESCRIPTION:
The aim of this study is to compare the accuracy of measuring the urea and creatinine level versus that of nitrazine test in vaginal wash of pre-labour rupture of membranes patients.Each patient with rupture of membranes will be assessed clinically and then if not in labour , patients will be divided into 2 groups, 5ml saline will be injected in the vagina of each patient in every group then the vaginal wash will be collected in a test tube. Urea and creatinine group, biochemical tests for urea and creatinine in mIU/ml to detect their presence in the wash will be done. In Nitrazine group wash will be assessed by nitrazine paper showing bluish discoloration in rupture membranes. Sensitivity of each test in diagnosed rupture of membranes will be assessed.Which means how many patients in each test show positive results in case of diagnosed case.

ELIGIBILITY:
Inclusion Criteria:

* Gestational age between 28 and 41 weeks
* Single intrauterine pregnancy
* History of gush of fluid
* Liquor detected on speculum examination

Exclusion Criteria:

* Vaginal bleeding
* Patients in labour
* Contaminated samples

Ages: 30 Years to 40 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 105 (Estimated)
Dates: Start 2014-05; Primary Completion 2021-12 (Estimated); Study Completion 2021-12 (Estimated)

PRIMARY OUTCOMES:
Urea and creatinine in vaginal fluid | Within first 24 hours after rupture of membranes in third trimester
  5ml saline will be injected vaginally then vaginal fluid will be collected.

SECONDARY OUTCOMES:
Nitrazine test | Within first 24 hours after rupture of membranes in third trimester
  5ml saline is injected vaginally then vaginal fluid is collected

CONTACTS AND LOCATIONS:
Overall Officials: Nesreen A Shehata, MD, Principal Investigator — Beni-Suef University
Locations (1):
- Nesreen Abdel Fattah Abdullah Shehata, Cairo, Egypt